CLINICAL TRIAL: NCT06639256
Title: An Open-label, Multiple-center, Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of HY07121 Powder for Solution for Infusion in Patients With Advanced Solid Tumors
Brief Title: Phase 1/2 Clinical Study of HY07121 Powder for Solution for Infusion in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HY0007-101
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Safety; Tolerability; Efficacy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product HY07121 for Dose Escalation (Experimental): PART ONE- Dose escalation: HY07121 should be administered intravenously at recommended dose. The purpose of the Dose Escalation Phase (Part one) is to characterize the safety and tolerability of the test product HY07121 and determine the maximum tolerated dose (MTD) (if any) and/or the recommended dose(s) (RD) based on the frequency of the occurrence of Dose-Limiting Toxicity (DLT) in each cohort during the DLT evaluation period.
  Interventions: Drug: Test Product HY07121
- Test product HY07121 for Dose Expansion (Experimental): PART TWO- Dose expansion: HY07121 should be administered intravenously at recommended dose. Patients will be administered a recommended dose of HY07121 established from the Dose Escalation Phase of the study.
  Interventions: Drug: Test Product HY07121

INTERVENTIONS:
Drug: Test Product HY07121 — HY07121 should be administered intravenously at recommended dose.
  Other Names: HY0007-101

SUMMARY:
This is a multi-center, open-label, phase 1/2 study to evaluate the safety, efficacy, and pharmacokinetic (PK)/pharmacodynamic (PD) characteristics of HY07121 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The study starts with a dose escalation part (Part 1) followed by a dose expansion part (Part 2). The main purpose of this study is to evaluate the safety and tolerability of the drug HY07121 and determine the maximum tolerated dose (MTD) (if any) and/or the recommended dose(s) (RD) and preliminary anti-tumor activity. Additional purposes of the study are to evaluate the pharmacokinetics (PK) properties, immunogenicity, correlation of the biomarkers and PK profile with anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* ≥18 years old and ≤80 years old, gender: male or female;
* Histologically or cytologically confirmed unresectable advanced/metastatic solid tumor that has relapsed or progressed on or after standard systemic treatments, or refused the standard treatment, or for which no standard treatment is available;
* Presence of at least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status score is 0 or 1;
* Life expectancy ≥3 months;
* Participant must have adequate main organ function;
* Fertile female patients must have a negative serological pregnancy test within 7 days before the first dosing and be willing to use effective birth control/contraception to prevent pregnancy during the study period up to 6 months after the last dosing of the study. Male patients must agree to have no sperm donation plans and to use effective contraceptive methods during the study period until 6 months after the last dose of the study. Postmenopausal women must have amenorrhea for at least 12 months before they are considered infertile.

Exclusion Criteria:

* Within the defined washout periods for prior anti-cancer treatments;
* Participant is currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of first dose of HY07121.
* Any other malignancy within 2 years prior to the first dose of the study treatment except for localized cancers that are considered to have been cured and in the opinion of the Investigator present a low risk for recurrence.
* Participant has not recovered (i.e., to Grade 1 or to baseline) from previous anticancer therapy-induced Adverse Events (AEs).
* Participants with a history of recently (within previous 2 years of the first dose of the study treatment) active diverticulitis or symptomatic peptic ulcer disease;
* Major surgery within 4 weeks of receiving the first dose of study treatment;
* Participant has Symptomatic Central Nervous System (CNS) metastases, or CNS metastases requiring CNS-directed local therapy (such as radiotherapy or surgery) or corticosteroids therapy within 4 weeks of first dose of study treatment;
* Participants with untreated or under treatment for tuberculosis, including but not limited to tuberculosis; Patients who have received standardized anti-tuberculosis treatment and have been confirmed cured by the researchers can be included;
* Participants with clinically significant cardiovascular diseases, in the past 6 months prior to the first dose of the study treatment; symptomatic coronary heart disease requiring drug treatment; arrhythmia requiring drug treatment; or uncontrolled hypertension;
* Known Human Immunodeficiency Virus (HIV) infection or known Acquired Immunodeficiency Syndrome (AIDS);
* Active or chronic hepatitis B or hepatitis C infection; treponema pallidum antibody positive, and confirmed positive test;
* Active known or suspected autoimmune disease.
* History of non-infectious pneumonitis that has required a course of oral or intravenous steroids to assist with recovery, or interstitial lung disease or severe obstructive pulmonary disease;
* History of severe allergy;
* History of allogeneic organ transplantation or graft-versus-host disease;
* Have received live/attenuated vaccines and mRNA vaccines within 4 weeks prior to screening or plan to receive live/attenuated vaccines and mRNA vaccines during the study period;
* Any active infection requires systemic treatment via intravenous infusion within 4 weeks prior to the first dose of study treatment;
* Known psychiatric disorder or drug abuse that would interfere the trial requirements;
* Participant with uncontrolled pleural effusion, pericardial effusion or peritoneal effusion or need drainage;
* In addition to the tumors present at the time of entry into the study, other active malignancies were present within 3 years prior to the first dose (not excluding locally cured tumors, such as skin basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the breast, etc.);
* Participants considered unsuitable for participation in this study by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation (Part One): Incidence and Nature of Dose-Limiting Toxicity (DLT) | 21 days during the first 3-week cycle
  Dose-Limiting Toxicity (DLT) will be defined using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or American Society for Transplantation and Cellular Therapy (ASTCT) criteria for Cytokine Release Syndrome (CRS).
Dose Escalation (Part One): Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | Up to 2 years
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
Dose Escalation (Part One): Percentage of participants experiencing Adverse Event (AE) related dose interruptions, dose delays, and dose intensity | Up to 2 years
  Occurrence of Adverse Event (AE) related dose interruptions, dose delays and dose intensity (duration of HY07121 exposure)
Dose Expansion (Part Two): Objective Response Rate (ORR) | Up to 2 years
  Proportion of participants who have a confirmed Complete Response (CR) or a Partial Response (PR)

SECONDARY OUTCOMES:
Dose Expansion (Part Two): Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | Up to 2 years
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
Dose Expansion (Part Two): Percentage of participants experiencing adverse event (AE) related dose interruptions, dose delays, and dose intensity | Up to 2 years
  Occurrence of adverse event (AE) related dose interruptions, dose delays and dose intensity (duration of HY07121 exposure).
Dose Escalation and Expansion: Assessment of HY07121 Cmax | Up to 2 years
  Maximum concentration observed (Cmax) observed from the pharmacokinetic profile
Dose Escalation and Expansion: Assessment of HY07121 AUC | Up to 2 years
  Area under the concentration versus time curve calculated using the trapezoidal method
Dose Escalation and Expansion: Assessment of HY07121 T1/2 | Up to 2 years
  The time it takes for half the drug concentration to be eliminated calculated using slope of the terminal line
Dose Escalation and Expansion: Assessment of HY07121 anti-drug-antibody (ADA) | Up to 2 years
  Incidence, duration, titer of serum anti-HY07121 antibody (ADA)
Dose Escalation (Part One): Objective Response Rate (ORR) | Up to 2 years
  Proportion of participants who have a confirmed complete response (CR) or a Partial Response (PR) determined by Investigator per the Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1
Dose Escalation and Expansion: Duration Of Response (DOR) assessed by investigator per Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 | Up to 2 years
  Duration Of Response (DOR) is defined as the time from the measurement criteria are first met for complete response (CR) /Partial Response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease.
Dose Escalation and Expansion: Disease Control Rate (DCR) assessed by investigator per RECIST Version 1.1 | Up to 2 years
  Disease Control Rate is defined as the percentage of participants who have achieved CR or PR or have demonstrated stable disease
Dose Escalation and Expansion: Progression-Free Survival (PFS) assessed by investigator per RECIST Version 1.1 | Up to 2 years
  Progression-Free Survival (PFS) is defined as the time from the date of first administration of HY07121 to the date of the first documented disease progression determined by Investigator as per RECIST 1.1 or death from any cause, whichever occurs first
Dose Escalation and Expansion: Time-To-Progression (TTP) assessed by investigator per RECIST Version 1.1 | Up to 2 years
  Time-To-Progression (TTP) is defined as the time from the date of first administration of HY07121 to the date of the first documented disease progression
Dose Escalation and Expansion: Overall Survival (OS) | Up to 2 years
  Overall Survival (OS) is defined as the time from the date of first administration of HY07121 to death due to any cause
Dose Escalation and Expansion: The correlation between tumor biomarkers and efficacy | Up to 2 years
  Objective Response Rate (ORR) is defined as proportion of participants who have a confirmed Complete Response (CR) or a Partial Response (PR) determined by Investigator per RECIST version 1.1. Tumor biomarkers will be tested using Immunohistochemistry (IHC) and scored using Tumor Proportion Score (TPS) and/or Combined Positive Score (CPS) algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Huiyura666! Yu, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Cancer Hospital of Shandong First Medical University, Jinan, China